CLINICAL TRIAL: NCT04951843
Title: The Effect of Black Soybeans Koji Product Supplementation on Nutrients Absorption and Anti-aging Effect in Elderly
Brief Title: Koji Product Supplementation' s Study
Acronym: KPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201806058RINA
Record Dates: First submitted 2019-04-15; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Sarcopenia
Keywords: protein
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Black soybean koji product (Experimental): Oral supplement 2 servings of black soybean koji product per day, for 10 weeks.
  Interventions: Dietary Supplement: Black soybean koji product

INTERVENTIONS:
Dietary Supplement: Black soybean koji product — Black soybean koji product

SUMMARY:
The present project is to identify the effect of black soy beans Koji product supplementation on nutrients absorption and anti-aging effect in elderly.

DETAILED DESCRIPTION:
Previous studies show that supplementation of soy protein can effectively increase muscle mass and protein utilization. Besides, soy extracts and isoflavones can stimulate muscle growth by activating the anabolic pathway of muscle tubules. Black soybean is known to be rich in legume protein and isoflavones.We speculate that black soybean supplementation can improve the nutritional status and muscle mass of elderly people, thereby delaying the deterioration of muscular dystrophy in the elderly. Reduce the occurrence of debilitation in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* 1-2 items are necessary, 3-5 can match one item

  1. Age above 65 years
  2. Oral intake
  3. Walking speed: ≤ 0.8 m/s (measured by time for a 5-meter usual gait)
  4. Handgrip strength: Men: <26 kg Women: <18 kg (measured by electronic hand grip dynamometer)
  5. Calf circumference: Men: ≤ 34 cm Women: ≤ 33 cm

Exclusion Criteria:

1. Participant in a moderate or strenuous exercise
2. Unable to walk
3. Unable to take in food from the mouth
4. People who can't record or communicate.
5. Refuse to accept the 3-day diet record
6. Allergic to black soybeans or legumes
7. Allergic to egg or milk
8. Infected with disease and had to be hospitalized for treatment before 4 weeks of the intervention test start
9. A patient who has been diagnosed with a malignant tumor or has a history of malignancy in the past year.
10. The estimated glomerular filtration rate (eGFR) is less than 60 ml/min/1.73 m2 in the past three months.
11. Hypothyroidism
12. People who often have symptoms of gastrointestinal upset.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Body mass index | Change from baseline outcome measure at 10th week (post-test)
  Measure Participants' detected body composition by using bioelectrical impedance analysis (BIA) as a non-invasive test instrument to measure body mass index (BMI).
Fat mass | Change from baseline outcome measure at 10th week (post-test).
  Measure Participants' detected body composition by using bioelectrical impedance analysis (BIA) as a non-invasive test instrument to measure fat mass.
Muscle mas | Change from baseline outcome measure at 10th week (post-test)
  Measure Participants' detected body composition by using bioelectrical impedance analysis (BIA) as a non-invasive test instrument to measure whole body and appendicular skeletal muscle mass.
Visceral fat area(VFA) | Change from baseline outcome measure at 10th week (post-test)
  Measure Participants' detected body composition by using bioelectrical impedance analysis (BIA) as a non-invasive test instrument to measure Visceral fat area(VFA) (cm2).
BIA - Basal Metabolic Rate(BMR) | Change from baseline outcome measure at 10th week (post-test)
  Measure Participants' detected body composition by using bioelectrical impedance analysis (BIA) as a non-invasive test instrument to measure Basal Metabolic Rate(BMR) (kcal)
  .
whole body Mineral | Change from baseline outcome measure at 10th week (post-test)
  Measure Participants' detected body composition by using bioelectrical impedance analysis (BIA) as a non-invasive test instrument to measure Mineral (kg) in whole body.
  .
Bone Mineral Content | Change from baseline outcome measure at 10th week (post-test)
  Measure Participants' detected body composition by using bioelectrical impedance analysis (BIA) as a non-invasive test instrument to measure Bone Mineral Content (kg).
Cellular Water | Change from baseline outcome measure at 10th week (post-test)
  Measure Participants' detected body composition by using bioelectrical impedance analysis (BIA) as a non-invasive test instrument to measure whole body Extracellular Water (L), Intracellular Water(L), and Total Body Water (L), et al.
  .
Muscle Strength - Hand Grip Strength | Change from baseline outcome measure at 10th week (post-test)
  Using hand grips to measure hand grip strength.
Physical Performance - Walking Speed | Change from baseline outcome measure at 10th week (post-test)
  Measuring participants' speed to walk 5 ft.
Gut Microbiota Composition Analysis | Change from baseline outcome measure at 10th week (post-test)
  Total genome DNA from samples was extracted from stool samples using the CTAB/SDS method. One hundred ng of DNA was amplified with barcoded primers16S V3+V4: 314F-806R annealing to the V3-V4region of the 16S rRNA. All of the PCR reactions were carried out using a Phusion® High-Fidelity PCR Master Mix (New England Biolabs, Location). Samples with a bright main strip between 400 and 450bp were selected from 2% agarose gel for further experiments. Mixture PCR products were purified using a Qiagen Gel Extraction Kit (Qiagen, Germany). Libraries were generated with the TruSeq® DNA PCR-Free Sample Preparation Kit and quantified with Qubit and Q-PCR. The purified DNA was then sequenced using the HiSeq2500 PE250 (Company, Location).
Gut Microbiota -derived Metabolite Analysis | Change from baseline outcome measure at 10th week (post-test)
  Measurements of short-chain fatty acids in feces during the experiment by using gas chromatography.
Inflammatory Cytokines TNF-α Analysis | Change from baseline outcome measure at 10th week (post-test)
  The inflammation-associated serum cytokines TNF-α was analyzed using colorimetric kits (Company, Location). Thioredoxin (Cloud-Clone Corp, SEA702Hu, City, State, USA) and Complement Component 5a (Cloud-Clone Corp, SEA388Hu) in the urine was evaluated for the effects of inflammation states and also assessed using colorimetric kits. The procedures followed the kit instructions and were measured using an ELISA reader (Bio Tek, PowerWave XS2, City, State, USA).
Inflammatory Cytokines IL-6 Analysis | Change from baseline outcome measure at 10th week (post-test)
  The inflammation-associated serum cytokines IL-6 was analyzed using colorimetric kits (Company, Location). Thioredoxin (Cloud-Clone Corp, SEA702Hu, City, State, USA) and Complement Component 5a (Cloud-Clone Corp, SEA388Hu) in the urine was evaluated for the effects of inflammation states and also assessed using colorimetric kits. The procedures followed the kit instructions and were measured using an ELISA reader (Bio Tek, PowerWave XS2, City, State, USA).
Inflammatory Cytokines IL-1β Analysis | Change from baseline outcome measure at 10th week (post-test)
  The inflammation-associated serum cytokines IL-1β (BioLegend, City, State, USA) was analyzed using colorimetric kits (Company, Location). Thioredoxin (Cloud-Clone Corp, SEA702Hu, City, State, USA) and Complement Component 5a (Cloud-Clone Corp, SEA388Hu) in the urine was evaluated for the effects of inflammation states and also assessed using colorimetric kits. The procedures followed the kit instructions and were measured using an ELISA reader (Bio Tek, PowerWave XS2, City, State, USA).
Red blood cells analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of red blood cells( M/ul)
Hemoglobin analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of Hemoglobin(g/dL).
MCHC(g/dL) analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of MCHC(g/dL)
Albumin analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of albumin(g/dL).
Hematocrit analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of Hematocrit(%).
RDW-CV analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of RDW-CV(%).
HbA1C analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of HbA1C(%).
MCV analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of MCV(fL).
MCH analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of MCH(pg).
Platelets analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of Platelets(k/uL).
WBC analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of WBC(k/uL) .
AST analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of AST(U/L).
ALT analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of ALT(U/L).
GGT analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of GGT(U/L).
T-Cholesterol analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of T-Cholesterol(mg/dL).
Triglyceride analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of triglyceride(mg/dL).
BUN analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of BUN(mg/dL).
Uric acid analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of Uric acid(mg/dL).
HDL-C analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of HDL-C(mg/dL).
LDL-C analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of LDL-C(mg/dL).
hs-CRP analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of hs-CRP(mg/dL).
Fasting blood glucose analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of fasting blood glucose(mg/dL).
Creatinine analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of creatinine(mg/dL).
Free T4 analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of 【Free T4(ng/dL)】
hsTSH analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of 【hsTSH(ulU/dL)】
HOMA-IR analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of 【 HOMA-IR】
Insulin analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of 【 insulin(uU/dL)】
eGFR analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of 【eGFR (mL/min/1.73^2)】
Ca analysis | Change from baseline outcome measure at 10th week (post-test)
  Use the Clinical Chemistry Analyzer to detection of Ca(mmol/dL).
specific gravity index analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes specific gravity index (USG).
Urine pH analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes pH.
Urine total protein analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes Total protein (mg/dL).
Urine glucose analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes glucose (-/+).
Urine Urea Nitrogen analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes Urine Urea Nitrogen(-/+).
Urine ketones analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes ketones(-/+).
Urine Creatinine analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes Creatinine(mg/dL).
Urine bilirubin (dipstick) analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes bilirubin (-/+).
Urine Albumin analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes Albumin(mg/L).
Urine Albumin/Creatinine analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes Albumin/Creatinine(mg/g).
Urine Nitrite (dipstick) analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes Nitrite(-/+).
Urine WBC esterase analysis | Change from baseline outcome measure at 10th week (post-test)
  Fasting for 8 hours, collecting 10ml urine. Routine urine analysis which includes WBC esterase(-/+).
Superoxide dismutase (SOD) Oxidative stress assessment | Change from baseline outcome measure at 10th week (post-test)
  Oxidative stress assessment to assess Superoxide dismutase (SOD) in serum was measured by the ELISA kit.
Glutathione peroxidase (GPx) Oxidative stress assessment | Change from baseline outcome measure at 10th week (post-test)
  Oxidative stress assessment to assess Glutathione peroxidase (GPx) in serum was measured by the ELISA kit..
Catalase Oxidative stress assessment | Change from baseline outcome measure at 10th week (post-test)
  Oxidative stress assessment to assess Catalase in serum was measured by the ELISA kit..
Physical examination-Height | Change from baseline outcome measure at 10th week (post-test)
  Measure participants' height. The height measurement method is to measure after you take off your shoes and step on the machine.
Physical examination- Body weight | Change from baseline outcome measure at 10th week (post-test)
  Measure participants' body weight. The body weight measurement method is to measure after you take off your shoes and step on the weight machine.
Physical examination - waist circumference | Change from baseline outcome measure at 10th week (post-test)
  Measure participants' waist circumference. The waist measurement method is to use a tape measure to measure the waist circumference above the human hips.
Physical examination - arm circumference | Change from baseline outcome measure at 10th week (post-test)
  Measure participants' arm circumference. The measurement method of the arm circumference is the circumference of the upper arm and is measured at the mid-point between the tips of the shoulder and elbow. .
Physical examination - calf circumference | Change from baseline outcome measure at 10th week (post-test)
  Measure participants' calf circumference. The measurement method of the calf circumference should be the same as the shoulder width and place the tape measure at the thickest part of the calf with a horizontal line around it for measurement.
Physical examination - hip circumference | Change from baseline outcome measure at 10th week (post-test)
  Measure participants' hip circumference. The hip measurement method is to use a tape measure to measure the maximum hip diameter.

SECONDARY OUTCOMES:
Physical Activity Questionnaire assessment | Change from baseline outcome measure at 10th week (post-test)
  Using Physical Activity Questionnaire to assess participants' activity level.
24-hour Dietary Recall Form | Change from baseline outcome measure at 10th week (post-test)
  The 24-hour diet recall method is conducted by interviewers who have received professional training in food serving size. Ask participants to recall all food and beverages actually consumed in the past 24 hours and record them in the questionnaire. Location, and the name, material, quantity and preparation method of food; among them, the estimation of the quantity can be assisted by using food weighing tools and food quantitative aids.
Gastrointestinal Function Assessment | Change from baseline outcome measure at 10th week (post-test)
  Assess the number of bowel movements, bowel habits, bowel pattern, and flatulence
Mini nutrition assessment | Change from baseline outcome measure at 10th week (post-test)
  This Mini nutrition assessment is a Indicator of nutrition status .The score range from 0-30,24 to 30 points represent Normal nutritional status, 17 to 23.5 points represent At the risk of malnutrition, less than 17 points represent Malnourished.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Yu Huang, Ph.D, Study Chair — Taipei Medical University Graduate Institute of Metabolism and Obesity Sciences
Locations (1):
- Taipei Medical University, Taipei, Taiwan